CLINICAL TRIAL: NCT01696630
Title: Phase II Study, Randomized, Monocentric, Single-blind, Comparing the Efficacy of Xenon and Desflurane, in Association With a Thoracic Epidural Analgesia in the Maintenance Phase of a Colorectal Oncologic Surgery
Brief Title: Xenon Combined With Intraoperative Thoracic Epidural Analgesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: XENON; 2012-002155-41 (EudraCT Number); ET2012-19 (Other: Sponsor's number)
Record Dates: First submitted 2012-09-21; First posted 2012-10-01 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: anesthesia, epidural anagesia, colorectal surgery, xenon, hemodynamic change
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Xenon; Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desflurane (Active Comparator): Desflurane 6.5% (+/-0.5%) in association with a thoracic epidural analgesia in maintenance phase
  Interventions: Drug: Desflurane
- Xenon (Experimental): Xenon 60% (+/-5%) in association with a thoracic epidural analgesia in maintenance phase
  Interventions: Drug: Xenon

INTERVENTIONS:
Drug: Xenon
  Arms: Xenon
Drug: Desflurane
  Arms: Desflurane

SUMMARY:
This is a monocentric study in 2 steps: A safety part to assess the feasibility of using Xenon in association with a thoracic epidural analgesia (TEA) with a sequential recruitment of 3, 6 or 9 patients according to predefined safety rules. The second part will randomly allocated patients (1:1) to receive TEA+Xenon or TEA+Desflurane. 28 patients will be enrolled and followed over 45 days.

DETAILED DESCRIPTION:
The first step is divided into 3 parts. 9 patients will be sequentially enrolled (3 patients in each part). The patients will be followed during 45 days and the following rules will be used to assess the safety:

First part: if no toxicity: initiation of the randomised part. If 1/3 toxicity: start of the second part. If 2 or 3/3 toxicity: end of the study.

Second part: same rules and possible start of the third part. Third part: if no toxicity: initiation of the randomised part. If 1 or more toxicity: end of the study.

The safety will be assessed after each part by an independent data safety monitoring board.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Planned surgery for oncologic colic and/or rectal surgery
* ASA score I or II
* Indication of complementary thoracic epidural analgesia
* Agree to use an effective form of contraception
* Patients who can understand, read and write French language
* Covered by a medical insurance
* Patients who have dated/signed an inform consent

Exclusion Criteria:

* Unstable angina within the 30 last days
* Myocardial infarction within 28 days prior to surgery
* Uncontrolled arterial high blood pressure
* Severe cardiac insufficiency
* Severe chronic obstructive pneumopathy
* Patient who requires FiO2 > 40%
* Patient already enrolled in a clinical study which may interfere with the present study
* Known hypersensitivity to one of the study drugs
* History or familial history of malignant hyperthermia
* Documented high intracranial pressure
* Eclampsia or pre-eclampsia
* Pregnant or breastfeeding woman
* Liver injury (icterus) and/or unexplained fever and/or eosinophilia after halogen exposure
* Failure in epidural anesthesia installation
* Patient refusal
* Patient who can't be compliant to the present protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Variation of intraoperative Mean Arterial Pressure (MAP) | Maintenance phase
  Variation between the Mean Arterial Pressure (MAP) at induction and the mean of intraoperative MAP values in each patient and comparaison between arms.

SECONDARY OUTCOMES:
Measure of hemodynamic parameters (Systolic Ejection Volume, Heart rate, DeltaPP) | Throughout the maintenance of anesthesia, an expected average of 6 hours
  monitoring device (automatic recorder)
Delay from the surgery to the discharge date | from the surgery to the hospital discharge date
  Delay from the date of surgery to the date of hospital discharge (days)
Delay between the end of surgery and Post Anesthesia Care Unit's exit (min) | from the end of surgery up to Post Anesthesia Care Unit's exit
  Delay between the end of surgery and Post Anesthesia Care Unit's exit (min)
Total dose requirement of Vasopressive and hypotensive agents | Throughout the maintenance of anesthesia, an expected average of 6 hours
Volume of each product infused | Throughout the maintenance of anesthesia, an expected average of 6 hours
Total dose of morphine | Throughout the maintenance of anesthesia, an expected average of 6 hours
  Total dose of morphine required to maintain BIS between 40 and 60 (in mg/kg)
Quality of awaking | 5 minutes after eyes opening
  Modified Aldrete score and Recovery Index
Delay to oral feeding recovery | From surgery to oral feeding reintroduction
  Time from the date of surgery to the date of first subsequent oral food intake
Post-operative Adverse Events | 45 days after surgery
  Post-operative Adverse Events (according to the NCI-CTC version 4.03)
post-operative pain | At entrance and exit of post operative room and 24 hours after the end of anesthesia
  Score to Visual Analog Scale
Delay to intestinal transit recovery | Time to postoperative stools
  Time from the date of surgery to the date of first postoperative stools

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, France

REFERENCES:
- [Background] Nakata Y, Goto T, Ishiguro Y, Terui K, Kawakami H, Santo M, Niimi Y, Morita S. Minimum alveolar concentration (MAC) of xenon with sevoflurane in humans. Anesthesiology. 2001 Apr;94(4):611-4. doi: 10.1097/00000542-200104000-00014. PMID 11379681
- [Background] Rasmussen LS, Schmehl W, Jakobsson J. Comparison of xenon with propofol for supplementary general anaesthesia for knee replacement: a randomized study. Br J Anaesth. 2006 Aug;97(2):154-9. doi: 10.1093/bja/ael141. Epub 2006 Jun 17. PMID 16782975
- [Background] Salmi E, Laitio RM, Aalto S, Maksimow AT, Langsjo JW, Kaisti KK, Aantaa R, Oikonen V, Metsahonkala L, Nagren K, Korpi ER, Scheinin H. Xenon does not affect gamma-aminobutyric acid type A receptor binding in humans. Anesth Analg. 2008 Jan;106(1):129-34, table of contents. doi: 10.1213/01.ane.0000287658.14763.13. PMID 18165567
- [Background] CULLEN SC, GROSS EG. The anesthetic properties of xenon in animals and human beings, with additional observations on krypton. Science. 1951 May 18;113(2942):580-2. doi: 10.1126/science.113.2942.580. No abstract available. PMID 14834873
- [Background] Wappler F, Rossaint R, Baumert J, Scholz J, Tonner PH, van Aken H, Berendes E, Klein J, Gommers D, Hammerle A, Franke A, Hofmann T, Schulte Esch J; Xenon Multicenter Study Research Group. Multicenter randomized comparison of xenon and isoflurane on left ventricular function in patients undergoing elective surgery. Anesthesiology. 2007 Mar;106(3):463-71. doi: 10.1097/00000542-200703000-00010. PMID 17325504
- [Background] Baumert JH, Hein M, Hecker KE, Satlow S, Schnoor J, Rossaint R. Autonomic cardiac control with xenon anaesthesia in patients at cardiovascular risk. Br J Anaesth. 2007 Jun;98(6):722-7. doi: 10.1093/bja/aem083. Epub 2007 Apr 27. PMID 17468494
- [Background] Luttropp HH, Thomasson R, Dahm S, Persson J, Werner O. Clinical experience with minimal flow xenon anesthesia. Acta Anaesthesiol Scand. 1994 Feb;38(2):121-5. doi: 10.1111/j.1399-6576.1994.tb03852.x. PMID 7909641
- [Background] Rossaint R, Reyle-Hahn M, Schulte Am Esch J, Scholz J, Scherpereel P, Vallet B, Giunta F, Del Turco M, Erdmann W, Tenbrinck R, Hammerle AF, Nagele P; Xenon Study Group. Multicenter randomized comparison of the efficacy and safety of xenon and isoflurane in patients undergoing elective surgery. Anesthesiology. 2003 Jan;98(1):6-13. doi: 10.1097/00000542-200301000-00005. PMID 12502972
- [Background] Dupont J, Tavernier B, Ghosez Y, Durinck L, Thevenot A, Moktadir-Chalons N, Ruyffelaere-Moises L, Declerck N, Scherpereel P. Recovery after anaesthesia for pulmonary surgery: desflurane, sevoflurane and isoflurane. Br J Anaesth. 1999 Mar;82(3):355-9. doi: 10.1093/bja/82.3.355. PMID 10434815
- [Background] Stuttmann R, Jakubetz J, Schultz K, Schafer C, Langer S, Ullmann U, Hilbert P. Recovery index, attentiveness and state of memory after xenon or isoflurane anaesthesia: a randomized controlled trial. BMC Anesthesiol. 2010 May 7;10:5. doi: 10.1186/1471-2253-10-5. PMID 20459661
- [Background] Diemunsch P; Societe francaise d'anesthesie et de reanimation. [Conference of experts--short text. Management of postoperative nausea and vomiting. French Society of Anesthesia and Resuscitation]. Ann Fr Anesth Reanim. 2008 Oct;27(10):866-78. doi: 10.1016/j.annfar.2008.09.004. Epub 2008 Oct 25. No abstract available. French. PMID 18952398